CLINICAL TRIAL: NCT02347748
Title: The Impact of Comfort Talk on Anxiety Levels and Procedural Experience in a Pediatric Population Undergoing Cardiac Catheterization: A Prospective Randomized Controlled Trial
Brief Title: Comfort Talk for Pediatric Cardiac Catheterization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Jacqueline Viegas, RN, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 1000046792
Record Dates: First submitted 2015-01-21; First posted 2015-01-27 (Estimated); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Anxiety; Pain; Adaptation, Psychological; Stress, Psychological
Keywords: Pain; Anesthesia Recovery Period; Postoperative Period; Adaptation, Psychological; Relaxation; Stress, Psychological
MeSH Terms: conditions — Anxiety Disorders; Pain; Stress, Psychological

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group A - Reading pre-procedure script (Experimental): Patients will be read a pre-procedure comfort talk script in the pre-procedure work-up area
  Interventions: Behavioral: Reading pre-procedure script
- Group B - Reading pre-extubation script (Experimental): Patients will be read a pre-extubation script;
  Interventions: Behavioral: Reading pre-extubation script
- Group C - Reading 2 scripts (Experimental): Patients will be read a pre-procedure comfort talk script in the pre-procedure work-up area Patients will be read a pre-extubation script
  Interventions: Behavioral: Reading pre-procedure script; Behavioral: Reading pre-extubation script; Behavioral: Reading 2 scripts
- Group D (No Intervention): Patients will not be read any script

INTERVENTIONS:
Behavioral: Reading pre-procedure script — Patients will be read a pre-procedure comfort talk script in the pre-procedure work-up area
  Arms: Group A - Reading pre-procedure script; Group C - Reading 2 scripts
Behavioral: Reading pre-extubation script — Patients will be read a comfort talk script before extubation
  Arms: Group B - Reading pre-extubation script; Group C - Reading 2 scripts
Behavioral: Reading 2 scripts — Patients will be read a pre-procedure comfort talk script in the pre-procedure work-up area.
  Patients will be read a comfort talk script before extubation
  Arms: Group C - Reading 2 scripts

SUMMARY:
Background: Pre anaesthesia anxiety in children is a strong predictor of postoperative behavior challenges and outcomes. In addition, intra-operative stress can precipitate post-traumatic stress symptomatology. Comfort Talk, consisting of rapport, relaxation, and reframing of potentially stressful experiences, applied pre-operatively in script form, has been highly successful in alleviating anxiety and positively affecting procedural outcomes in adult patients undergoing interventional procedures. No published literature exists evaluating its' impact in paediatric cardiac catheterization. Purpose: To investigate the impact of comfort talk on the level of pre-induction anxiety, procedural and recovery experience, as well as short-term post-procedural behaviour and satisfaction after discharge in pediatric patients undergoing cardiac catheterization procedures. Design: Prospective randomized, double blind controlled trial. Participants: 160 children, ages 7-18 years, having a cardiac catheterization procedure under general anaesthesia. Intervention: Group A will be read a pre-procedure comfort talk script in the pre-procedure work-up area; Group B will be read a pre-extubation (before the breathing tube is removed) script ; Group C will be read a pre-procedure plus a pre-extubation script; Group D will not be read any script. All groups will be treated according to the standard of care approaches usually provided for anaesthesia, catheterization, and recovery. Outcomes: We will compare the effect of the script strategy on preoperative anxiety. Procedural and recovery measurements will include room time in the catheterization suite, time to discharge from the recovery room; drug use, vomiting, rebleeds, and cardiorespiratory stability. Postoperative behaviour will be assessed by questionnaire. Postoperative anxiety and pain will be secondary outcome measures using queries on 0-10 verbal self-report scales Hypotheses are:

1. Patients being read a preoperative Comfort Talk script will experience less anxiety prior to anaesthesia induction.
2. The reduction of anxiety prior to induction is associated with better immediate and short-term recovery outcomes.
3. Patients being read a pre-extubation script will recover better than controls.
4. The combination of a pre-procedure script and a pre-extubation script will have the greatest positive effect on physical and emotional well-being in the immediate recovery period and at short term follow-up.

DETAILED DESCRIPTION:
Among scheduled children for cardiac catheterization at the Labatt Family Health Center Cardiac Diagnostic and Interventional Unit (CDIU) , potential participants will be identified at their pre-catheterization clinic visit, the study explained, and informed consent obtained. On the day of their procedure, participants will be randomized to one of 4 groups. In the pre-catheterization work-up area, a modified Yale Preoperative Anxiety Scale (mYPAS) plus anxiety and pain self-ratings on verbal 0-10 scales will be obtained. In intervention groups A and C a pre-procedure Comfort Talk script will be read while the parent or guardian is present. Patients in Group B and D will not have a script read. The participants will be reassessed by mYPAS and asked to rate their level of pain and anxiety again on entering the procedure room and then care will continue as usual. The team members and anaesthesiologist will be blinded to the prior treatment and behave naturally but abstain from formalized use of hypnosis, invitation to imagery, use of scripts or electronic means of distraction. Induction of anaesthesia and the procedure will continue according to laboratory routine. Use of premedication will be permitted as per judgement of the anaesthesiologist. After induction a Paediatric Anesthesia Behaviour score (PAB) rating will be obtained. Prior to extubation, one of the CDIU nurses will read the pre-extubation script for those subjects in Groups B and C. Extubation and transfer to recovery will follow usual routine.

When the patients are transferred to the recovery room nurses will be unaware of group attribution. On waking from anaesthesia and up to 6 hours post-operatively, participants will again be asked to rate their levels of pain and anxiety at various intervals.

Within 24-48 hours of discharge from the hospital, families will be called to follow-up on their experience in the CDIU using the follow-up questionnaire regularly used by the CDIU nurses. At the same time the parents will be reminded to fill in the Post Hospitalization Behaviour Questionnaire (PHBQ) reflecting the child's behaviour in the first week after the procedure and mail it back in the stamped addressed envelope provided. If the envelope has not been mailed back within 10 days one of the research team members will call and complete it with the parents over the phone.

The pre-procedure script is based on a script that three large prospective randomized trials found to be effective in adults in reducing anxiety, pain, and complications of invasive image-guided procedures. It has been modified for use in paediatrics. The standardized script containing relaxing and hypnoidal language with suggestions for coping strategies will be read by CDIU RNs trained in Comfort Talk in the pre-catheterization work-up area. The pre-extubation script contains suggestions for healing, recovery, functioning of bodily systems, and acknowledgement of the patient's contribution.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for cardiac catheterization
* Procedure performed under general anesthetic
* Ability to speak and understand English
* No apparent cognitive impairments

Exclusion Criteria:

* Active dissociative psychiatric disease

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 160 (Actual)
Dates: Start 2015-01; Primary Completion 2018-06 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Pre-anesthesia Anxiety | 3-15 min prior to anesthesia induction
  Anxiety is measured by the modified Yale Preoperative Anxiety Scale (mYPAS) immediately upon entry into the operating room and introduction of the anesthesia mask to the child. The mYPAS consists of 22 items in five categories (activity, emotional expressivity, state of arousal, vocalization, and use of parents) and a maximal score of 100.
Postoperative Behavior | 1 week postoperatively
  Measured with the Post Hospitalization Behaviour Questionnaire (PHBQ)

SECONDARY OUTCOMES:
Satisfaction with care | 24-48 hrs after discharge from the hospital
  CDIU Post Cardiac Catherization follow-up phone survey addressing presence or absence of discomfort, bruising at the cath site, fever, return to normal bodily functions and activity, satisfaction with treatment from and communication with staff.
Procedure Time | Duration of the cardiac catheterization procedure (1-4 hrs depending on complexity of case)
  Duration of the cardiac catheterization procedure (1-4 hrs depending on complexity of case)
Recovery room time | within 24 hrs of procedure
  Measure per recovery room log
Drug usage during procedure | 1-4 hrs
  Amount of anesthesia drugs given in drug units
Drug usage during recovery | within 24 hrs
  Amount of sedatives and narcotics in drug units
Antiemetics | within 28 hrs
  Amount of antiememtics in drug units
Anesthesia induction behavior | within1 hr of anesthesia induction
  Measured by the Pediatric Anesthesia Behaviour Score (PAB)
Nausea | within 28 hrs of procedure start
  measured by frequency and severity
Rebleeds | within 1 week of procedure
  counts and severy
any pain | within 28 hrs of arrival
  0-10 self-reporting scale
Self-reported anxiety | within 28 hrs of arrival
  0-10 self-reporting scale

CONTACTS AND LOCATIONS:
Overall Officials: Jacquie Viegas, RN, Principal Investigator — Hospital for Sick Childen, Toronto, CA
Locations (1):
- Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Background] Kain ZN, Mayes LC, Cicchetti DV, Bagnall AL, Finley JD, Hofstadter MB. The Yale Preoperative Anxiety Scale: how does it compare with a "gold standard"? Anesth Analg. 1997 Oct;85(4):783-8. doi: 10.1097/00000539-199710000-00012. PMID 9322455
- [Background] Varughese AM, Nick TG, Gunter J, Wang Y, Kurth CD. Factors predictive of poor behavioral compliance during inhaled induction in children. Anesth Analg. 2008 Aug;107(2):413-21. doi: 10.1213/ane.0b013e31817e616b. PMID 18633018
- [Background] Yip P, Middleton P, Cyna AM, Carlyle AV. Non-pharmacological interventions for assisting the induction of anaesthesia in children. Cochrane Database Syst Rev. 2009 Jul 8;(3):CD006447. doi: 10.1002/14651858.CD006447.pub2. PMID 19588390
- [Background] Karling M, Stenlund H, Hagglof B. Child behaviour after anaesthesia: associated risk factors. Acta Paediatr. 2007 May;96(5):740-7. doi: 10.1111/j.1651-2227.2007.00258.x. PMID 17462064
- [Background] Kain ZN, Wang SM, Mayes LC, Caramico LA, Hofstadter MB. Distress during the induction of anesthesia and postoperative behavioral outcomes. Anesth Analg. 1999 May;88(5):1042-7. doi: 10.1097/00000539-199905000-00013. PMID 10320165
- [Background] Watson AT, Visram A. Children's preoperative anxiety and postoperative behaviour. Paediatr Anaesth. 2003 Mar;13(3):188-204. doi: 10.1046/j.1460-9592.2003.00848.x. No abstract available. PMID 12641680
- [Background] Lang EV, Benotsch EG, Fick LJ, Lutgendorf S, Berbaum ML, Berbaum KS, Logan H, Spiegel D. Adjunctive non-pharmacological analgesia for invasive medical procedures: a randomised trial. Lancet. 2000 Apr 29;355(9214):1486-90. doi: 10.1016/S0140-6736(00)02162-0. PMID 10801169
- [Background] Lang EV, Berbaum KS, Faintuch S, Hatsiopoulou O, Halsey N, Li X, Berbaum ML, Laser E, Baum J. Adjunctive self-hypnotic relaxation for outpatient medical procedures: a prospective randomized trial with women undergoing large core breast biopsy. Pain. 2006 Dec 15;126(1-3):155-64. doi: 10.1016/j.pain.2006.06.035. Epub 2006 Sep 7. PMID 16959427
- [Background] Lang EV, Berbaum KS, Pauker SG, Faintuch S, Salazar GM, Lutgendorf S, Laser E, Logan H, Spiegel D. Beneficial effects of hypnosis and adverse effects of empathic attention during percutaneous tumor treatment: when being nice does not suffice. J Vasc Interv Radiol. 2008 Jun;19(6):897-905. doi: 10.1016/j.jvir.2008.01.027. Epub 2008 Mar 17. PMID 18503905
- [Background] Butler LD, Symons BK, Henderson SL, Shortliffe LD, Spiegel D. Hypnosis reduces distress and duration of an invasive medical procedure for children. Pediatrics. 2005 Jan;115(1):e77-85. doi: 10.1542/peds.2004-0818. PMID 15629969
- [Background] Lang EV, Rosen MP. Cost analysis of adjunct hypnosis with sedation during outpatient interventional radiologic procedures. Radiology. 2002 Feb;222(2):375-82. doi: 10.1148/radiol.2222010528. PMID 11818602
- [Background] Montgomery GH, David D, Winkel G, Silverstein JH, Bovbjerg DH. The effectiveness of adjunctive hypnosis with surgical patients: a meta-analysis. Anesth Analg. 2002 Jun;94(6):1639-45, table of contents. doi: 10.1097/00000539-200206000-00052. PMID 12032044
- [Background] Faymonville ME, Meurisse M, Fissette J. Hypnosedation: a valuable alternative to traditional anaesthetic techniques. Acta Chir Belg. 1999 Aug;99(4):141-6. PMID 10499382
- [Background] Flory N, Lang E. Practical hypnotic interventions during invasive cancer diagnosis and treatment. Hematol Oncol Clin North Am. 2008 Aug;22(4):709-25, ix. doi: 10.1016/j.hoc.2008.04.008. PMID 18638697
- [Background] Davidson AJ. Awareness, dreaming and unconscious memory formation during anaesthesia in children. Best Pract Res Clin Anaesthesiol. 2007 Sep;21(3):415-29. doi: 10.1016/j.bpa.2007.05.001. PMID 17900018
- [Background] Crandall M, Lammers C, Senders C, Savedra M, Braun JV. Initial validation of a numeric zero to ten scale to measure children's state anxiety. Anesth Analg. 2007 Nov;105(5):1250-3, table of contents. doi: 10.1213/01.ane.0000284700.59088.8b. PMID 17959951
- [Background] Bringuier S, Dadure C, Raux O, Dubois A, Picot MC, Capdevila X. The perioperative validity of the visual analog anxiety scale in children: a discriminant and useful instrument in routine clinical practice to optimize postoperative pain management. Anesth Analg. 2009 Sep;109(3):737-44. doi: 10.1213/ane.0b013e3181af00e4. PMID 19690240
- [Background] Vernon DT, Schulman JL, Foley JM. Changes in children's behavior after hospitalization. Some dimensions of response and their correlates. Am J Dis Child. 1966 Jun;111(6):581-93. doi: 10.1001/archpedi.1966.02090090053003. No abstract available. PMID 5939538
- [Background] Karling M, Stenlund H, Hagglof B. Behavioural changes after anaesthesia: validity and liability of the Post Hospitalization Behavior Questionnaire in a Swedish paediatric population. Acta Paediatr. 2006 Mar;95(3):340-6. doi: 10.1080/08035250500434751. PMID 16497646
- [Background] Beringer RM, Greenwood R, Kilpatrick N. Development and validation of the Pediatric Anesthesia Behavior score--an objective measure of behavior during induction of anesthesia. Paediatr Anaesth. 2014 Feb;24(2):196-200. doi: 10.1111/pan.12259. Epub 2013 Sep 19. PMID 24103068
- [Derived] Viegas J, Holtby H, Runeckles K, Lang EV. The Impact of Scripted Self-Hypnotic Relaxation on the Periprocedural Experience and Anesthesiologist Sedation Use in the Pediatric Cardiac Catheterization Suite: A Prospective Randomized Controlled Trial. J Pain Res. 2022 Oct 27;15:3447-3458. doi: 10.2147/JPR.S373608. eCollection 2022. PMID 36324867